CLINICAL TRIAL: NCT00131742
Title: A Phase III Randomized, Double Blind Trial of LdT (Telbivudine) Versus Lamivudine in Chinese Adults With Compensated Chronic Hepatitis B
Brief Title: Telbivudine Versus Lamivudine in Chinese Adults With Compensated Chronic Hepatitis B
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Novartis Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NV-02B-015
Record Dates: First submitted 2005-08-18; First posted 2005-08-19 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Telbivudine; Lamivudine

INTERVENTIONS:
Drug: telbivudine
Drug: lamivudine

SUMMARY:
This study is being conducted to compare the effectiveness and safety of telbivudine (LdT) and lamivudine in Chinese adults.

ELIGIBILITY:
Inclusion Criteria:

* Documented clinical history compatible with chronic hepatitis B infection

Other protocol-defined inclusion criteria may apply

Exclusion Criteria:

* Patient is pregnant or breastfeeding
* Patient is co-infected with hepatitis C virus (HCV), hepatitis D virus (HDV) or HIV
* Patient has previously received lamivudine or any investigational anti-HBV nucleoside or nucleotide analog

Other protocol-defined exclusion criteria may apply

Ages: 16 Years to 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Dates: Start 2004-07; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing, China

REFERENCES:
- [Derived] Hou J, Yin YK, Xu D, Tan D, Niu J, Zhou X, Wang Y, Zhu L, He Y, Ren H, Wan M, Chen C, Wu S, Chen Y, Xu J, Wang Q, Wei L, Chao G, Constance BF, Harb G, Brown NA, Jia J. Telbivudine versus lamivudine in Chinese patients with chronic hepatitis B: Results at 1 year of a randomized, double-blind trial. Hepatology. 2008 Feb;47(2):447-54. doi: 10.1002/hep.22075. PMID 18080339